CLINICAL TRIAL: NCT05781360
Title: A Phase I First-in-human, Open-label, Multicenter Study to Investigate the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of SIM0237 in Adult Participants with Advanced Solid Tumors
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of SIM0237 in Adult Participants with Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: An internal business decision, not based on safety or regulatory considerations.
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: Shanghai Xianxiang Medical Technology Co., Ltd. (Industry); Simcere Zaiming (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SIM0237-101
Record Dates: First submitted 2023-02-17; First posted 2023-03-23 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Locally Advanced Unresectable or Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: PART ONE- Dose escalation (Experimental): The purpose of the Dose Escalation Phase (Part one) is to characterize the safety and tolerability of SIM0237 and determine the maximum tolerated dose (MTD) (if any) and/or the recommended dose(s) (RD) based on the frequency of the occurrence of DLTs in each cohort during the DLT evaluation period.
  Interventions: Drug: SIM0237
- Experimental: PART TWO- Dose expansion (Experimental): Patients will be administered a recommended dose of SIM0237 established from the Dose Escalation Phase of the study.
  Interventions: Drug: SIM0237

INTERVENTIONS:
Drug: SIM0237 — SIM0237 should be administered intravenously at recommended dose qw or other dosing regimens

SUMMARY:
This is a multicenter, open-label, phase I study to evaluate the safety, efficacy, and pharmacokinetic (PK)/pharmacodynamic(PD) characteristics of SIM0237 in participants with advanced solid tumors.

DETAILED DESCRIPTION:
The study starts with a dose escalation part (Part 1) followed by a dose expansion part (Part 2). The main purpose of this study is to evaluate the safety and tolerability of SIM0237 and determine the maximum tolerated dose (MTD) (if any) and/or the recommended dose(s) (RD) and preliminary anti-tumor activity when given once every week or other dosing regimens. Additional purposes of the study are to evaluate the pharmacokinetics (PK) properties, immunogenicity, correlation of the biomarkers and PK profile with anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* ≥18 years of age;
* Histological/cytological diagnosis of selected locally advanced unresectable or metastatic solid tumor not amenable to local therapies (clinical diagnosis of HCC is allowed); participants must have failed to derive clinical benefit on standard therapies, or ineligible for the standard of care therapy
* Presence of at least one measurable lesion according to RECIST Version 1.1
* ECOG performance status score of 0 or 1;
* Life expectancy of ≥12 weeks;
* Participant must have adequate main organ function.
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 72 hours prior to the start of study treatment. WOCBP must be willing to use either 2 adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy or to abstain from heterosexual activity throughout the study, starting from the first dose of the study treatment through 180 days after the last dose of study treatment.
* Male participants must agree to use adequate contraception starting from the first dose of the study treatment through 180 days after the last dose of the study treatment.

Exclusion Criteria:

* Within the defined washout periods for prior anti-cancer treatments;
* Participant is currently participating or has participated in a study of an investigational agent or using an investigational device within 4 weeks of first dose of SIM0237.
* Any other malignancy within 2 years prior to the first dose of the study treatment except for localized cancers that are considered to have been cured and in the opinion of the Investigator present a low risk for recurrence.
* Participant has not recovered (i.e., to Grade 1 or to baseline) from previous anticancer therapy-induced AEs.
* Participants with a history of recently (within previous 2 years of the first dose of the study treatment) active diverticulitis or symptomatic peptic ulcer disease;
* Major surgery within 2 weeks of receiving the first dose of study treatment;
* Participant has symptomatic central nervous system (CNS) metastases, or CNS metastases requiring CNS-directed local therapy (such as radiotherapy or surgery) or corticosteroids therapy within 2 weeks of first dose of study treatment;
* Participants with a history of active pulmonary tuberculosis infection within 1 year; participants with history more than 1 year prior to the first dose of study treatment may be considered suitable if there is no evidence of active pulmonary tuberculosis judged by the Investigator;
* Participants with clinically significant cardiovascular diseases, in the past 6 months prior to the first dose of the study treatment; symptomatic coronary heart disease requiring drug treatment; arrhythmia requiring drug treatment; QTcF interval >480 msec; or uncontrolled hypertension;
* Participants who have ascites requiring drainage or pleural effusion or pericardial effusion requiring drainage within 28 days after previous drainage; Known human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS);
* Active or chronic hepatitis B or hepatitis C infection; participant with HBsAg positive or detective HBV-DNA at screening should receive antiviral treatment as per local practice during the study.
* Concomitant therapy with any other anti-cancer therapy or chronic use of immunosuppressive doses (more than 10 mg/day of prednisone or equivalent) of systemic corticosteroids.
* Active known or suspected autoimmune disease.
* History of non-infectious pneumonitis that has required a course of oral or intravenous steroids to assist with recovery, or interstitial lung disease or severe obstructive pulmonary disease;
* History of severe hypersensitivity reactions to mAbs;
* History of allogeneic organ transplantation or graft-versus-host disease;
* Use of any live vaccine therapy within 4 weeks prior to the first dose of study treatment;
* Any active infection requires systemic treatment via intravenous infusion within 2 weeks prior to the first dose of study treatment;
* Known psychiatric disorder or drug abuse that would interfere the trial requirements;
* Previous treatment with IL-15 agonists;
* Participant is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
* Other conditions that researchers consider inappropriate for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Dose Escalation (Part One): Incidence and nature of Dose-Limiting Toxicity (DLT) | 18 months
  DLTs will be defined using NCI CTCAE version 5.0 or ASTCT criteria for Cytokine Release Syndrome (CRS).
Dose Escalation (Part One): Percentage of participants experiencing treatment-emergent adverse events (TEAEs) | 18 months
  Incidence and severity of adverse events (AEs), serious adverse events (SAEs), and lab abnormalities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 and American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading
Dose Escalation (Part One): Percentage of participants experiencing AE related dose interruptions and dose delays, dose intensity | 18 months
  Occurrence of AE related dose interruptions, dose delays and dose intensity (duration of SIM0237 exposure).
Dose Expansion (Part Two): Objective Response Rate (ORR) | 12 months
  Proportion of participants who have a confirmed Complete Response (CR) or a Partial Response (PR), as the Best Overall Response (BOR) determined by Investigator per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Dose Expansion (Part Two): Percentage of participants experiencing treatment-emergent adverse events (TEAEs) | 18 months
  Incidence and severity of adverse events (AEs), serious adverse events (SAEs), and lab abnormalities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 and American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading
Dose Expansion (Part Two): Percentage of participants experiencing AE related dose interruptions and dose delays, dose intensity | 18 months
  Occurrence of AE related dose interruptions, dose delays and dose intensity (duration of SIM0237 exposure).
Dose Escalation and Expansion: Assessment of SIM0237 Cmax | 30 months
  Maximum concentration observed (Cmax) observed from the PK profile
Dose Escalation and Expansion: Assessment of SIM0237 AUC | 30 months
  Area under the concentration versus time curve calculated using the trapezoidal method
Dose Escalation and Expansion: Assessment of SIM0237 T1/2 | 30 months
  The time it takes for half the drug concentration to be eliminated calculated using slope of the terminal line
Dose Escalation and Expansion: Assessment of SIM0237 antibody (ADA) | 30 months
  Incidence, duration, titer of serum anti-SIM0237 ADA
Dose Escalation (Part One): Objective Response Rate (ORR) | 48 months
  Proportion of participants who have a confirmed complete response (CR) or a Partial Response (PR), as the Best Overall Response (BOR) determined by Investigator per the RECIST v1.1
Dose Escalation and Expansion: Duration Of Response (DOR) assessed by investigator per RECIST Version 1.1 | 48 months
  DOR is defined as the time from the measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease.
Dose Escalation and Expansion: Disease Control Rate (DCR) assessed by investigator per RECIST Version 1.1 | 48 months
  Disease Control Rate is defined as the percentage of participants who have achieved CR or PR or have demonstrated stable disease
Dose Escalation and Expansion: Progression-Free Survival (PFS) assessed by investigator per RECIST Version 1.1 | 48 months
  PFS is defined as the time from the date of first administration of SIM0237 to the date of the first documented disease progression determined by Investigator as per RECIST 1.1 or death from any cause, whichever occurs first
Dose Escalation and Expansion: Time-To-Progression (TTP) assessed by investigator per RECIST Version 1.1 | 48 months
  TTP is defined as the time from the date of first administration of SIM0237 to the date of the first documented disease progression
Dose Escalation and Expansion: Overall Survival (OS) | 48 months
  Overall Survival is defined as the time from the date of first administration of SIM0237 to death due to any cause
Dose Escalation and Expansion: ORR in participants with different PD-LI expression levels | 48 months
  ORR is defined as proportion of participants who have a confirmed Complete Response (CR) or a Partial Response (PR), as the Best Overall Response (BOR) determined by Investigator per RECIST v1.1. PD-L1 expression will be tested using 22C3 IHC and scored using TPS and/or CPS algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Bijoyesh Mookerjee, MD, Study Chair — Simcere Zaiming
Locations (9):
- United States (3):
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - NYU Langone, New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- China (6):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shandong Cancer Hospital, Jinan, Shandong
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang